CLINICAL TRIAL: NCT01524003
Title: Chinese Cancer Prevention Study(CHICAPS) Mass Population Based Cervical Cancer Screening
Brief Title: Chinese Cancer Prevention Study(CHICAPS)
Acronym: CHICAPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Preventive Oncology International, Inc. (Other)
Collaborators: Peking University Shenzhen Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CHICAPS
Record Dates: First submitted 2011-12-29; First posted 2012-02-01 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2015-05

CONDITIONS: Cervical Intraepithelial Neoplasia; Cervical Cancer; Cervical Neoplasm; Cervical Dysplasia; Human Papillomavirus
Keywords: community based participatory research
MeSH Terms: conditions — Uterine Cervical Dysplasia; Uterine Cervical Neoplasms | interventions — Cryotherapy; Colposcopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cryotherapy after VIA triage (Experimental): Women who test HPV positive will be randomized to the experimental arm or the standard of care arm. In the Experimental arm VIA will be done to determine acceptability for cryotherapy [R/O high-grade CIN too large for cryotherapy (usually 3-4 quadrant disease) or cancer]. All acceptable patients will have an ECC done and then immediate cryotherapy.
  Interventions: Procedure: cryotherapy
- Colposcopy and biopsy (Active Comparator): Standard of care. Women testing positive for HPV will be randomized to the experimental arm (immediate cryotherapy) or the Standard of care arm, for colposcopy, biopsy, and leep based on the pathology results.
  Interventions: Procedure: Colposcopy

INTERVENTIONS:
Procedure: cryotherapy — cryotherapy treatment of the uterine cervix
  Other Names: MedGyn cryotherapy; medical grade CO2
  Arms: Cryotherapy after VIA triage
Procedure: Colposcopy — Colposcopy, biopsy and LEEP based on the pathology results
  Other Names: Digital colposcopy; POI microbiopsy; LEEP
  Arms: Colposcopy and biopsy

SUMMARY:
The purpose of this study is to develop and implement a community based preventive healthcare model using cervical cancer screening as the target medical intervention.

The investigators will first conduct 2 pilot studies to refine their preventive healthcare model based on the principles of community based participatory research (1000 participants). The investigators will then apply the model to screen 9000 women for cervical cancer over a period of 7-9 days. This 10,000 patient trial will explore the ability of a community to conduct their own screening program to identify who needs medical intervention based on self-collection and centralized high-throughput low cost human papillomavirus (HPV) testing.

DETAILED DESCRIPTION:
Screening and prevention programs in general, throughout the world, suffer from major cost constraints, poor participation, lost to follow-up, and concerns about sustainability.

Over the past 15 years the investigators have been studying self-collection as a way to reach the medically underserved for cervical cancer screening. In a recent 10,000 patient randomized clinical trial they demonstrated that a self-collected sample is equivalent in accuracy to a physician obtained endocervical specimen and can be done less expensively and with higher throughput than all current and proposed accurate testing modalities.

With the majority of the worlds' medically underserved now living in middle income countries, it is no longer necessary to think small, slow, and simple, with poor quality control. It is totally achievable with self-collection to have centralized, high-throughput, low cost per case processing, and to reach millions of women in a short period of time. Again, these concepts need not be restricted to the medically underserved, but the clarity of this paradigm is a realistic solution for a critical developing world healthcare problem. In addition, we now have solid media specimen transport cards, thereby avoiding the logistics of dealing with personal use of alcohol-based liquids, concerns about exposure temperature, and ease of transportation. Using PCR-based technologies in a self-collection algorithm has the ability to not only make the testing highly sensitive, but help to address another key issue and that is how to manage the positives. In the investigators' proposed centralized model, since the primary output of the testing provides genotyping a reasonable option for tailoring the management of the positives would exist.

Now the need is to focus on developing the models that will enable them to efficiently place the existing technologies next to the women who need them the most. Developing community based systems that remove the identification of who is abnormal from the medical model, will markedly affect the cost of preventive healthcare. In addition with community involvement in the design of the program, it is expected that their participation in the "campaigns" and follow-up will be significantly improved. Sustainability also becomes a simpler problem because of the "campaign" or "event" type model (possibly once/year, or per every 5-10years). The investigators believe that the patient recruitment and loss to follow up observed in screening programs conducted in the developing world, have their roots in asking large numbers of patients, who are not presently ill, or symptomatic, to travel long distances and interrupt their daily life. The investigators believe that a much more effective program can be designed by the community, and using a self-collection model will ensure greater recruitment and participation, minimizing loss to follow up. This project CHICAPS is designed to further develop the community based screening model and in addition randomize treatment options to explore a technology more suited to rural environments

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria

1. Non pregnant women 35-59 years of age.
2. No hysterectomy
3. No prior pelvic radiation.
4. Willing to sign consent form

Exclusion Criteria:

1. Males
2. Women younger than 35 years old and older than 59 years old.
3. Pregnant women.
4. Patients with known history of hysterectomy or radiation for a pelvic cancer.
5. Refusal to participate

Ages: 35 Years to 59 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8382 (Actual)
Dates: Start 2011-11; Primary Completion 2013-07 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
The investigators will determine the percentage of the population in the target area that are reached by the screening protocol. | Ongoing for up to 36 months
  Pilot study will take up to 8 months. The community application will be complete approximately 5 months later and all follow up and data analysis will be complete in 36 months.
The investigators will determine the percentage of HPV screen positive women who return for evaluation and treatment. | Ongoing for up to 36 months
  Pilot study will take up to 8 months. The community application will be complete approximately 5 months later and all follow up and data analysis will be complete in 36 months

SECONDARY OUTCOMES:
The investigators will compare women treated in the standard of care arm and the experimental arm (VIA and cryotherapy) to determine the percentage of high grade disease at the 6 month follow-up and 2 year follow-up. | Ongoing for up to 36 months
  Pilot study will take up to 8 months. The community application will be complete approximately 5 months later and all follow up and data analysis will be complete in 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Jerome L Belinson, MD, Principal Investigator — Preventive Oncology International; Rufiang Wu, MD, Principal Investigator — Peking Universtiy Shenzhen Hospital
Locations (1):
- HeShan Public Health Department, Jiangmen Municipal City, Guangdong, China

REFERENCES:
- [Derived] Belinson JL, Wang G, Qu X, Du H, Shen J, Xu J, Zhong L, Yi J, Yi X, Wu R. The development and evaluation of a community based model for cervical cancer screening based on self-sampling. Gynecol Oncol. 2014 Mar;132(3):636-42. doi: 10.1016/j.ygyno.2014.01.006. Epub 2014 Jan 14. PMID 24440471